CLINICAL TRIAL: NCT04411056
Title: Time to Adapt in the Pandemic Era: A Prospective Randomized Study Comparing Time to Intubate With and Without the Barrier Box
Brief Title: A Study Comparing Time to Intubate With and Without a Barrier Box
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2004-38
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Intubation

STUDY DESIGN:
Intervention Model Description: Participants assigned to barrier box or no barrier box
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barrier box (Experimental): Participants will have a barrier box placed during intubation for a medical procedure. A barrier box is a medical device which was in use from May 1, 2020 to August 20, 2020 during the COVID-19 pandemic. The device is a barrier enclosure to protect healthcare providers caring for or performing medical procedures (such as intubation) on patients who are known or suspected to have COVID-19.
  Interventions: Other: Barrier box
- No Barrier box (No Intervention): Participants will have routine intubation with no barrier box

INTERVENTIONS:
Other: Barrier box — Placement of barrier box ( a plastic box for shielding)
  Arms: Barrier box

SUMMARY:
This study is for patients who will be having surgery and will have a breathing tube placed during intubation. The purpose of the research is to study the time it takes to use a barrier box for placement of a breathing tube. A barrier box is a clear box that sits over the head and shoulders of a patient as a breathing tube is placed. The box is used to protect the healthcare provider's exposure to coronavirus in patients who have COVID-19. The study will not include patients who test positive for COVID-19 or who are sick with COVID-19 symptoms. The researchers want to learn how long it takes to use the barrier box before it is used routinely in COVID-19 patients.

DETAILED DESCRIPTION:
The study will have two groups of 39 patients in each group. Some patients will have a barrier box and some patients will not have a barrier box. Patients will be randomly assigned to the barrier box or no barrier box group. The study will measure the time it takes to place the breathing tube.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting for surgery needing general anesthesia with endotracheal intubation
* pre-operatively tested negative for SARS- CoV-2 virus

Exclusion Criteria:

* inability to consent or cooperate,
* children
* pregnant women
* patients with severe cardiopulmonary compromise
* American Society Anesthesiologists' (ASA) physical status 4 and 5
* Body Mass Index (BMI) >35
* known or anticipated difficult airway
* patients with positive COVID status or unknown COVID status
* patients who reported claustrophobia in the pre-operative area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Praneeth Madabhushi, MD, MHCA, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Madabhushi P, Kinthala S, Ankam A, Chopra N, Porter BR. Time to adapt in the pandemic era: a prospective randomized non -inferiority study comparing time to intubate with and without the barrier box. BMC Anesthesiol. 2020 Sep 14;20(1):232. doi: 10.1186/s12871-020-01149-w. PMID 32928122
- See also: Publication PMID 32928122 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7488639/

RESULTS

PARTICIPANT FLOW:
Groups:
- Barrier Box: Participants will have a barrier box placed during intubation
  Barrier box: Placement of barrier box ( a plastic box for shielding)
Period: Overall Study
Arm/Group | Barrier Box | No Barrier Box
Started | 39 | 39
Completed | 38 | 38
Not Completed | 1 | 1
Not completed — surgery cancelled | 1 | 0
Not completed — Equipment problem during intubation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Barrier Box | No Barrier Box | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (16.7) | 52.7 (18.9) | 55.2 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 19 | 20 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38 | 38 | 76
American Society of Anesthesiology (ASA) Physical Status [Count of Participants; unit: Participants] — The American Society of Anesthesiology (ASA) Physical Status is used to assess a patient's pre-anesthesia medical condition and helps predict how patients will do during a surgical procedure. A lower ASA score predicts (but does not guarantee) better outcomes during a surgical procedure.
  * ASA 1 - a normal healthy patient
  * ASA 2 - a patient with mild systemic disease
  * ASA 3 - A patient with severe systemic disease.
  Participants
    ASA 1 | 1 | 2 | 3
    ASA 2 | 21 | 25 | 46
    ASA 3 | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubate
Description: Time to intubate refers to the time it takes to insert a tube into a patient's trachea to help them breathe. Intubation is a procedure routinely used before surgery to help keep the airway open. The study will compare the time to intubate in two groups, barrier box and no barrier box. In medical terms, time to intubate is the time from loss of twitches confirmed with a peripheral nerve stimulator to confirmation of end tidal carbon dioxide.
Time Frame: up to 2 minutes during intubation before surgery
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
seconds | 52.1 [26.1 to 78] | 42.0 [19.2 to 64.8]

2. Secondary Outcome: Intubation in First Attempt
Description: All participants were intubated successfully on the first attempt.
Time Frame: up to 2 minutes during intubation before surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
Participants | 38 | 38

3. Secondary Outcome: Need for Bag Mask Ventilation
Description: During induction time, there were no patients who needed bag mask ventilation. Bag mask ventilation is a technique used to provide oxygen and ventilation to patients who are not breathing adequately. Induction is the process of transitioning a patient from consciousness to unconsciousness at the beginning of a general anesthetic. The induction time is defined in medical terms as the time taken from propofol bolus to loss of twitches measured with a peripheral nerve stimulator.
Time Frame: up to 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
Participants | 0 | 0

4. Secondary Outcome: Participants' Lowest Blood Oxygen Level (Lowest Oxygen Saturation During Induction and Intubation)
Description: During process of inserting a tube in a patient's trachea (intubation) before surgery and the process of being given anesthesia (induction), there is a point where a patient's blood oxygen level drops to its lowest point during the process. This is referred to as the lowest oxygen saturation. In medical terms this is the lowest peripheral capillary oxygen saturation during the induction time defined as the time taken from propofol bolus to loss of twitches measured with a peripheral nerve stimulator.
  The maximum blood oxygen level is 100%. Normal range is 95% - 100%. Low oxygen level (hypoxemia)is below 95%.
Time Frame: up to 5 minutes
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
percentage of blood oxygen | 98.7 (2.6) | 98.8 (2.6)

5. Secondary Outcome: Induction Time
Description: Induction is the process of transitioning a patient from consciousness to unconsciousness at the beginning of a general anesthetic. The induction time is defined in medical terms as the time taken from propofol bolus to loss of twitches measured with a peripheral nerve stimulator.
Time Frame: up to 5 minutes
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
seconds | 65.9 [39.2 to 92.6] | 67.7 [43.7 to 91.7]

6. Other Pre Specified Outcome: Airway Assessment by Mallampati Score (Scale of 0 to 4)
Description: Airway assessment by Mallampati score (scale of 0 to 4) used to assess and prepare for possible difficult intubation of participants who score high. Lower scores are less likely to have a difficult intubation and higher scores are more likely to have a difficult intubation.
  Mallampati 0: Any part of the epiglottis is visible Mallampati 1: soft palate, uvula, and pillars are visible Mallampati 2: soft palate and uvula are visible Mallampati 3: only the soft palate and base of the uvula are visible Mallampati 4: only the hard palate is visible.
Time Frame: Up to 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
Participants
  Mallampati 0 | 0 | 0
  Mallampati 1 | 3 | 3
  Mallampati 2 | 29 | 31
  Mallampati 3 | 6 | 4
  Mallampati 4 | 0 | 0

7. Other Pre Specified Outcome: Airway Assessment by Thyromental Distance (TMD)
Description: Thyromental Distance (TMD) is the distance from the thyroid notch to the chin when the head is extended. TMD is used to assess and prepare for possible difficult intubation. A distance of greater than 3 finger breadth may be less likely to have a difficult intubation. A distance less than or equal to 3 finger breadth may be more likely to have a difficult intubation.
  Number of participants with TMD greater than 3 finger breadth will be assessed in both groups (Barrier Box and No Barrier Box).
Time Frame: Up to 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
Participants
  TMD greater than 3 finger breadth | 38 | 38
  TMD less than or equal to 3 finger breadth | 0 | 0

8. Other Pre Specified Outcome: Airway Assessment by Inter Incisor Distance
Description: Inter incisor distance is the distance between the upper and lower teeth of the open mouth of a patient. Inter incisor distance is used to assess and prepare for possible difficult intubation of participants who are less than or equal to 3 finger breadth. A distance greater than 3 finger breadth may be less likely to have a difficult airway or airway constriction.
  Number of participants with Inter incisor distance greater than 3 finger breadth will be assessed in both groups (Barrier Box and No Barrier Box).
Time Frame: Up to 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
Participants
  Inter incisor distance less than or equal to 3 finger breadth | 0 | 0
  Inter incisor distance greater than 3 finger breadth | 38 | 38

9. Other Pre Specified Outcome: Neck Range of Motion
Description: Neck range of motion is the degree of movement in the neck - how much the head can flex (bend forward), extend (tilt backwards), and rotate side to side. Neck range of motion helps assess and prepare for possible difficult intubation. Full range of motion is less likely for a difficult intubation. Restricted range of motion indicates a possible difficult intubation.
  Number of patients with Neck range of motion (categorized as full or restricted) will be assessed in both groups (Barrier Box and No Barrier Box)
Time Frame: Up to 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Barrier Box | No Barrier Box
Number analyzed (Participants) | 38 | 38
Participants
  Full | 36 | 38
  Restricted | 2 | 0

ADVERSE EVENTS:
Time Frame: One day during the surgery
Description: There were no deaths and no serious adverse events.
Arm/Group | Barrier Box | No Barrier Box
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT04411056/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT04411056/SAP_001.pdf